CLINICAL TRIAL: NCT03414944
Title: Elective Simultaneous Modulated Accelerated Brain Radiation Therapy for NSCLCs With Limited Brain Metastases,A Phase I,One-arm Trial
Brief Title: Elective Simultaneous Modulated Accelerated Brain Radiation Therapy for NSCLCs With Limited Brain Metastases
Acronym: SMART-Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, ShuanghuYuan, Director, Head of of Radiation Oncology, Principal Investigator, Clinical Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTOG1602
Record Dates: First submitted 2018-01-12; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Brain Metastases
Keywords: Non-small cell lung cancer; Brain metastases; SIB; hippocampus avoidance; inner ear avoidance
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART-Brain (Experimental): selective brain radiotherapy based on SIB and hippocampus, inner ear avoidance.
  Interventions: Radiation: SMART-Brain

INTERVENTIONS:
Radiation: SMART-Brain — Prescription dose: Gross tumor (PGTV) 40-50 Gy/10 fractions/2 weeks + EBI (PCTV) 30 Gy/10 fractions/2 weeks.
  OARs dose limits: Hippocampus D100%≤10Gy, Dmax≤17Gy,Inner ear: Dmean ≤15Gy.

SUMMARY:
Brain metastases are the most common intracranial tumors in adults. Whole-brain radiation therapy (WBI) increases the median survival of patients with brain metastases up to 3-6 months, but WBI can lead to the decline of cognition and quality of life, with short local control time. The use of SIB(simultaneous integrated boost) technology can increase the local control rate. Hippocampus avoidance can effectively reduce the cognitive impairment caused by WBI.This study was designed to evaluate the safety and efficacy of selective brain radiotherapy (EBI)(based on SIB and hippocampus, inner ear avoidance )in NSCLCs with limited brain metastases.

DETAILED DESCRIPTION:
In this prospective phase 1 study evaluating the safety and efficacy of selective brain radiotherapy in NSCLCs with limited brain metastases, patients will received selective brain radiotherapy based on SIB and hippocampus, inner ear avoidance.

Prescription dose: Gross tumor (PGTV) 40-50 Gy/10 fractions/2 weeks + EBI (PCTV) 30 Gy/10 fractions/2 weeks.

OARs dose limits: Hippocampus D100%≤10Gy, Dmax≤17Gy,Inner ear: Dmean ≤15Gy. All patients were observed and recorded daily for acute radiation impairment during radiotherapy. Follow-up every 2 months will be performed after radiotherapy.

The primary endpoint:Acute and chronic radiation response, QOL in patients, vestibular function,neurocognitive function based on mini-mental state examination(MMSE) questionnaires, hearing.

The secondary endpoint included:objective response rate (ORR);intracranial progression-free survival (iPFS); OS (defined as the time from study beginning to death from any cause).

ELIGIBILITY:
Inclusion Criteria:

histologically or cytologically confirmed NSCLC with MRI confirmed new brain metastases a life expectancy of at least 3 months; adequate organ function according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0.

Exclusion Criteria:

radiologically or pathologically confirmed metastases in the spinal cord or meninges obvious hernia formation risk previously received brain surgery or radiotherapy a history or presence of poorly controlled systemic diseases pregnant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12-02 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
AE | up to 12 months
  Adverse events

SECONDARY OUTCOMES:
iPFS | From date of treatment begining until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Intracranial progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shuanghu, doctor, Study Chair — Shandong cancer hospital and constitute
Locations (1):
- Shandong Cancer Hospital, Jin'an, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Result] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Result] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Result] Meyers CA, Brown PD. Role and relevance of neurocognitive assessment in clinical trials of patients with CNS tumors. J Clin Oncol. 2006 Mar 10;24(8):1305-9. doi: 10.1200/JCO.2005.04.6086. PMID 16525186
- [Result] Meyers CA, Smith JA, Bezjak A, Mehta MP, Liebmann J, Illidge T, Kunkler I, Caudrelier JM, Eisenberg PD, Meerwaldt J, Siemers R, Carrie C, Gaspar LE, Curran W, Phan SC, Miller RA, Renschler MF. Neurocognitive function and progression in patients with brain metastases treated with whole-brain radiation and motexafin gadolinium: results of a randomized phase III trial. J Clin Oncol. 2004 Jan 1;22(1):157-65. doi: 10.1200/JCO.2004.05.128. PMID 14701778
- [Result] Miller JA, Kotecha R, Suh JH. Comparative effectiveness of stereotactic radiosurgery versus whole-brain radiation therapy for patients with brain metastases from breast or non-small cell lung cancer. Cancer. 2016 Oct 15;122(20):3243-3244. doi: 10.1002/cncr.30188. Epub 2016 Jul 8. No abstract available. PMID 27392066
- [Result] Ozdemir Y, Yildirim BA, Topkan E. Whole brain radiotherapy in management of non-small-cell lung carcinoma associated leptomeningeal carcinomatosis: evaluation of prognostic factors. J Neurooncol. 2016 Sep;129(2):329-35. doi: 10.1007/s11060-016-2179-9. Epub 2016 Jun 15. PMID 27306442
- [Result] Mekhail T, Sombeck M, Sollaccio R. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. Curr Oncol Rep. 2011 Aug;13(4):255-8. doi: 10.1007/s11912-011-0180-1. No abstract available. PMID 21584645
- [Derived] Jiang A, Sun W, Zhao F, Wu Z, Shang D, Yu Q, Wang S, Zhu J, Yang F, Yuan S. Dosimetric evaluation of four whole brain radiation therapy approaches with hippocampus and inner ear avoidance and simultaneous integrated boost for limited brain metastases. Radiat Oncol. 2019 Mar 15;14(1):46. doi: 10.1186/s13014-019-1255-7. PMID 30876444